CLINICAL TRIAL: NCT03014609
Title: Cardiovascular Risk and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Cardiovascular Risk and Chronic Obstructive Pulmonary Disease
Acronym: ECO-COPD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.245
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; cardiovascular risk; inflammation; oxidative stress; peripheral muscle function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be collected for each patient at the inclusion visit and follow-up visits. Parameters of inflammation, cardiovascular risk, oxidative stress and metabolic function will be measured.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The principal objective of the study is to measure parameters of inflammation, oxidative stress, and vascular, respiratory, and peripheral muscle function parameters, and identify parameters indicative of evolving cardiovascular risk (CVR) in COPD patients, using multivariate analysis.

DETAILED DESCRIPTION:
Reduced lung function is a major risk factor for cardiovascular mortality (CV), regardless of age, sex and history of smoking. Similarly, CV events are known causes of mortality in patients with chronic obstructive pulmonary disease (COPD). The investigators propose to determine the parameters influencing the evolution of CV risk in a cohort of COPD patients followed over 5 years. For this the investigators will study the role of inflammation, oxidative stress, and vascular, respiratory and peripheral muscle function parameters.

In order to study a sufficient number of patients the investigators propose to group data from two cohorts: a first cohort of 121 COPD patients that already exists (currently closed to inclusions but still undergoing follow-up (NCT00404430)) and a new cohort of 150, decompensated or not, COPD patients.

This study is of major scientific interest and will enable to obtain extremely important information to better understand COPD.

ELIGIBILITY:
Inclusion Criteria:

For patients with stable COPD:

* Men or women aged 18 to 85
* FEV1/FVC < 70% or proven BPCO
* Patients who have given their free and informed consent in writing

For patients with decompensated COPD:

* Men or women aged 18 to 85
* FEV1/FVC < 70% or proven BPCO
* At the time of acute respiratory failure (ARF), when admitted to hospital:

  * Respiratory rate > 25 cycles per minute
  * PaCO2 > 45 mmHg
  * blood pH < 7.35
* When included in the study:

  * pH > 7.33 at the end of ARF, 2 days in a row, or 3 to 7 days post-D1 decompensation (admission to the hospital)
  * Fever < 38.5°C
* Patients who have given their free and informed consent in writing

Exclusion Criteria:

* Obvious evolving infection or CRP > 100 mg/L
* Cardiac decompensation considered the main cause of decompensation or chronic heart failure with LVEF < 45%
* Evolving neoplasia
* On antioxidants: N-acetyl-cysteine, selenium, vit. C, vit. E
* Pregnant or nursing women
* Patients under tutorship or curatorship
* Patients participating in a drug clinical research study
* Patients not affiliated to the French social security system (or equivalent)
* Patients deprived of liberty or hospitalized without consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD Patients will be recruited during the consultations in Pneumology Department or in the Laboratory of Sleep (patients with stable COPD) or during their hospitalization in Medical Reanimation Unit (patients with decompensated COPD) at the University Grenoble Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change of the pulse wave velocity (PWV) | During 5 years since inclusion (once a year)
  Measurement of pulse wave velocity (PWV), which reflects cardiovascular risk (CVR).
  This measure will be performed at each visit (V1, V1 bis, V2, V3, V4, V5 and V6).

SECONDARY OUTCOMES:
Monitoring of COPD exacerbations compared to evolution of PWV | During 5 years since inclusion
  Determination of the relationship between exacerbations and the evolution of the PWV.
Relationship between the new cardiovascular (CV) events and the evolution of the PWV. | During 5 years since inclusion (once a year)
  Follow-up of exacerbations compared to new CV events (including myocardial infarction with or without ST segment elevation, ischemic stroke, unexplained sudden death at 5 years).
Correlations between the parameters of severity of pulmonary disease and physical activity. | During 5 years since inclusion (once a year)
  Measurement of extent of pulmonary disease; exploration of peripheral muscle function; measurement of physical activity; measurements of endothelial function; measurement of cardiac function.
Prevalence of nocturnal "non-dipping" of blood pressure during COPD. | During 5 years since inclusion (once a year)
  Measurement of ambulatory arterial blood pressure during 24 hours
Impact of sleep disorders and sleep apnea syndrome on the evolution of CVR during COPD. | At inclusion visit
  Measurement of sleep disorders and Sleep Apnea Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, ProfessorPHD, Principal Investigator — University Grenoble Hospital
Locations (1):
- University Grenoble Hospital, Grenoble, La Tronche, France

REFERENCES:
- [Result] Gan WQ, Man SF, Senthilselvan A, Sin DD. Association between chronic obstructive pulmonary disease and systemic inflammation: a systematic review and a meta-analysis. Thorax. 2004 Jul;59(7):574-80. doi: 10.1136/thx.2003.019588. PMID 15223864
- [Result] Mallia P, Johnston SL. Mechanisms and experimental models of chronic obstructive pulmonary disease exacerbations. Proc Am Thorac Soc. 2005;2(4):361-6; discussion 371-2. doi: 10.1513/pats.200504-025SR. PMID 16267363
- [Result] de Torres JP, Cordoba-Lanus E, Lopez-Aguilar C, Muros de Fuentes M, Montejo de Garcini A, Aguirre-Jaime A, Celli BR, Casanova C. C-reactive protein levels and clinically important predictive outcomes in stable COPD patients. Eur Respir J. 2006 May;27(5):902-7. doi: 10.1183/09031936.06.00109605. Epub 2006 Feb 2. PMID 16455829
- [Result] Malo O, Sauleda J, Busquets X, Miralles C, Agusti AG, Noguera A. [Systemic inflammation during exacerbations of chronic obstructive pulmonary disease]. Arch Bronconeumol. 2002 Apr;38(4):172-6. Spanish. PMID 11953269
- [Result] Dekhuijzen PN, Aben KK, Dekker I, Aarts LP, Wielders PL, van Herwaarden CL, Bast A. Increased exhalation of hydrogen peroxide in patients with stable and unstable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):813-6. doi: 10.1164/ajrccm.154.3.8810624.
- [Result] Rahman I. The role of oxidative stress in the pathogenesis of COPD: implications for therapy. Treat Respir Med. 2005;4(3):175-200. doi: 10.2165/00151829-200504030-00003. PMID 15987234
- [Result] Heunks LM, Vina J, van Herwaarden CL, Folgering HT, Gimeno A, Dekhuijzen PN. Xanthine oxidase is involved in exercise-induced oxidative stress in chronic obstructive pulmonary disease. Am J Physiol. 1999 Dec;277(6):R1697-704. doi: 10.1152/ajpregu.1999.277.6.R1697. PMID 10600916
- [Result] Yende S, Waterer GW, Tolley EA, Newman AB, Bauer DC, Taaffe DR, Jensen R, Crapo R, Rubin S, Nevitt M, Simonsick EM, Satterfield S, Harris T, Kritchevsky SB. Inflammatory markers are associated with ventilatory limitation and muscle dysfunction in obstructive lung disease in well functioning elderly subjects. Thorax. 2006 Jan;61(1):10-6. doi: 10.1136/thx.2004.034181. Epub 2005 Nov 11. PMID 16284220
- [Result] Carter R, Holiday DB, Nwasuruba C, Stocks J, Grothues C, Tiep B. 6-minute walk work for assessment of functional capacity in patients with COPD. Chest. 2003 May;123(5):1408-15. doi: 10.1378/chest.123.5.1408. PMID 12740255
- [Result] Mador MJ, Kufel TJ, Pineda LA, Sharma GK. Diaphragmatic fatigue and high-intensity exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 Jan;161(1):118-23. doi: 10.1164/ajrccm.161.1.9903010. PMID 10619807
- [Result] Saey D, Debigare R, LeBlanc P, Mador MJ, Cote CH, Jobin J, Maltais F. Contractile leg fatigue after cycle exercise: a factor limiting exercise in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2003 Aug 15;168(4):425-30. doi: 10.1164/rccm.200208-856OC. Epub 2003 Apr 24. PMID 12714348
- [Result] Engelen MP, Schols AM, Does JD, Wouters EF. Skeletal muscle weakness is associated with wasting of extremity fat-free mass but not with airflow obstruction in patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2000 Mar;71(3):733-8. doi: 10.1093/ajcn/71.3.733. PMID 10702166
- [Result] Barreiro E, de la Puente B, Minguella J, Corominas JM, Serrano S, Hussain SN, Gea J. Oxidative stress and respiratory muscle dysfunction in severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 15;171(10):1116-24. doi: 10.1164/rccm.200407-887OC. Epub 2005 Feb 25. PMID 15735057
- [Result] Debigare R, Cote CH, Maltais F. Peripheral muscle wasting in chronic obstructive pulmonary disease. Clinical relevance and mechanisms. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1712-7. doi: 10.1164/ajrccm.164.9.2104035. No abstract available. PMID 11719314
- [Result] Heunks LM, Dekhuijzen PN. Respiratory muscle function and free radicals: from cell to COPD. Thorax. 2000 Aug;55(8):704-16. doi: 10.1136/thorax.55.8.704. No abstract available. PMID 10899251
- [Result] Hunninghake DB. Cardiovascular disease in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2005;2(1):44-9. doi: 10.1513/pats.200410-050SF. PMID 16113468
- [Result] Rennard SI. Clinical approach to patients with chronic obstructive pulmonary disease and cardiovascular disease. Proc Am Thorac Soc. 2005;2(1):94-100. doi: 10.1513/pats.200410-051SF. PMID 16113475
- [Result] Gan WQ, Man SF, Sin DD. The interactions between cigarette smoking and reduced lung function on systemic inflammation. Chest. 2005 Feb;127(2):558-64. doi: 10.1378/chest.127.2.558. PMID 15705996
- [Result] MacCallum PK. Markers of hemostasis and systemic inflammation in heart disease and atherosclerosis in smokers. Proc Am Thorac Soc. 2005;2(1):34-43. doi: 10.1513/pats.200406-036MS. PMID 16113467
- [Result] Vassilakopoulos T, Karatza MH, Katsaounou P, Kollintza A, Zakynthinos S, Roussos C. Antioxidants attenuate the plasma cytokine response to exercise in humans. J Appl Physiol (1985). 2003 Mar;94(3):1025-32. doi: 10.1152/japplphysiol.00735.2002. Epub 2002 Nov 27. PMID 12571133
- [Result] Lerman A, Zeiher AM. Endothelial function: cardiac events. Circulation. 2005 Jan 25;111(3):363-8. doi: 10.1161/01.CIR.0000153339.27064.14. No abstract available. PMID 15668353
- [Result] Vivodtzev I, Minet C, Wuyam B, Borel JC, Vottero G, Monneret D, Baguet JP, Levy P, Pepin JL. Significant improvement in arterial stiffness after endurance training in patients with COPD. Chest. 2010 Mar;137(3):585-92. doi: 10.1378/chest.09-1437. Epub 2009 Oct 31. PMID 19880908
- [Result] Minet C, Vivodtzev I, Tamisier R, Arbib F, Wuyam B, Timsit JF, Monneret D, Borel JC, Baguet JP, Levy P, Pepin JL. Reduced six-minute walking distance, high fat-free-mass index and hypercapnia are associated with endothelial dysfunction in COPD. Respir Physiol Neurobiol. 2012 Aug 15;183(2):128-34. doi: 10.1016/j.resp.2012.06.017. Epub 2012 Jun 18. PMID 22721944
- [Result] Vivodtzev I, Tamisier R, Baguet JP, Borel JC, Levy P, Pepin JL. Arterial stiffness in COPD. Chest. 2014 Apr;145(4):861-875. doi: 10.1378/chest.13-1809. PMID 24687708
- [Result] Weidemann F, Herrmann S, Stork S, Niemann M, Frantz S, Lange V, Beer M, Gattenlohner S, Voelker W, Ertl G, Strotmann JM. Impact of myocardial fibrosis in patients with symptomatic severe aortic stenosis. Circulation. 2009 Aug 18;120(7):577-84. doi: 10.1161/CIRCULATIONAHA.108.847772. Epub 2009 Aug 3. PMID 19652094
- [Result] Marin JM, Soriano JB, Carrizo SJ, Boldova A, Celli BR. Outcomes in patients with chronic obstructive pulmonary disease and obstructive sleep apnea: the overlap syndrome. Am J Respir Crit Care Med. 2010 Aug 1;182(3):325-31. doi: 10.1164/rccm.200912-1869OC. Epub 2010 Apr 8. PMID 20378728
- [Result] Vivodtzev I, Minet C, Tamisier R, Arbib F, Borel JC, Baguet JP, Levy P, Pepin JL. Arterial stiffness by pulse wave velocity in COPD: reliability and reproducibility. Eur Respir J. 2013 Oct;42(4):1140-2. doi: 10.1183/09031936.00014813. No abstract available. PMID 24081763
- [Result] Patel AR, Kowlessar BS, Donaldson GC, Mackay AJ, Singh R, George SN, Garcha DS, Wedzicha JA, Hurst JR. Cardiovascular risk, myocardial injury, and exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Nov 1;188(9):1091-9. doi: 10.1164/rccm.201306-1170OC. PMID 24033321
- [Result] Labarere J, Renaud B, Fine MJ. How to derive and validate clinical prediction models for use in intensive care medicine. Intensive Care Med. 2014 Apr;40(4):513-27. doi: 10.1007/s00134-014-3227-6. Epub 2014 Feb 26. PMID 24570265